CLINICAL TRIAL: NCT04273607
Title: Anticoagulation-free VV ECMO for Acute Respiratory Failure: A Pilot Safety and Feasibility Randomized Clinical Trial
Brief Title: Anticoagulation-free VV ECMO for Acute Respiratory Failure
Acronym: A-FREE ECMO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Damian Ratano (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor-Investigator, Damian Ratano, Principal Investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-5692.0
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: Extracorporeal membrane oxygenation; Anticoagulation; Thrombosis; Hemorrhage
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No anticoagulation (Experimental): Participants in this arm will not receive unfractionated heparin during the course of ECMO. They will receive standard venous thromboembolism prophylaxis with subcutaneous enoxaparin or unfractionated heparin
  Interventions: Drug: Subcutaneous Heparin
- Anticoagulation, ECMO standard of care (No Intervention): Participants in this arm will receive the standard of care anticoagulation with unfractionated heparin during the course of ECMO.

INTERVENTIONS:
Drug: Subcutaneous Heparin — The intervention group will receive prophylactic heparin instead of standard of care therapeutic intravenous heparin
  Other Names: Enoxaparin or unfractionated heparin
  Arms: No anticoagulation

SUMMARY:
Currently international experts recommend therapeutic anticoagulation for veno-venous extracorporeal membrane oxygenation (VV-ECMO). Reports and case series suggest that the absence of therapeutic anticoagulation is safe for VV-ECMO. No randomized control trials have assessed this. The aim of this pilot study is to assess safety and feasibility of an "anticoagulation-free strategy" for veno-venous ECMO (VV-ECMO) in Acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Although anticoagulation targets and monitoring strategies vary around the world, the current practice is still to anticoagulate patients on ECMO, mostly with UFH. However, the use of heparin coated circuits has changed their thrombogenicity. Preliminary data suggest that a low-dose unfractionated heparin (UFH) strategy is non-inferior to a therapeutic dose UFH. Indeed, in daily practice, when a patient on ECMO has severe bleeding complications, UFH is often stopped until the hemorrhagic issue is under control, sometimes for days. This has led some to hypothesize that anticoagulation might not be necessary for VV-ECMO, and a few case series report little to no increase in adverse events as a result. There are currently no randomized controlled trials comparing anticoagulation to no anticoagulation for patients supported with ECMO. Anticoagulation is, for physiological reasons, less necessary during VV-ECMO than VA-ECMO and this is the reason why our pilot study will focus on VV-ECMO only. Whereas the whole ECMO device is identical for both configurations, the risk of systemic embolization (e.g., stroke) and its severe complications is much higher in VA-ECMO where blood is reinjected directly into the systemic arterial system. Moreover, in the presence of severely decreased left ventricular function requiring VA-ECMO, the risk of left ventricular thrombus is very high and requires anticoagulation. During VV-ECMO, the risk of systemic embolization is low because the whole circuit is on the right side of the heart and relatively preserved biventricular function is needed to perform VV-ECMO

The hypothesis is that VV-ECMO is safe and feasible without therapeutic anticoagulation for adults with ARDS.

The objectives of this study is to assess, through a pilot study, the safety and feasibility of an "anticoagulation free strategy" for veno-venous ECMO (VV-ECMO) in acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with ARDS on VV-ECMO

Exclusion Criteria:

* Contraindication to anticoagulation with UFH (known heparin-induced thrombocytopenia, active hemorrhage, any surgery precluding the use of anticoagulation),
* Indication for therapeutic anticoagulation (pulmonary embolism or deep vein thrombosis, chronic anticoagulation therapy before ECMO insertion)
* Low-flow (<2 liters/min) VV-ECMO (ECCO2R)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
ECMO associated thrombotic complications | through ECMO completion, an average of 14 days
  Composite outcome of:
  * ECMO membrane oxygenator function assessed by trans-membrane pressure drop (> 10mmHg/l/min) and a membrane PaO2/FiO2 ratio (< 200mmHg)
    * Need to change ECMO circuit due to clotting or dysfunction
    * Platelets drop >50% in 24 hours and <50 /mm3
    * Development of a clinically significant thromboembolic event
  * Clinical deep vein thrombosis, clinically suspected and confirmed by ultrasound
  * Acute ischemic stroke, clinically suspected and confirmed by head-CT

SECONDARY OUTCOMES:
Hemorrhagic complications | through ECMO completion, an average of 14 days
  Hemorrhagic complications assessed and adapted as per Bleeding Academic Research Consortium (BARC)
  * Type 0: No bleeding
  * Type 1: Bleeding requiring transfusion of packed red blood cells (PRBC) or reduction of UFH
  * Type 2: Bleeding requiring transfusion of PRBC and reduction of UFH
  * Type 3: Life-threatening bleeding requiring, transfusion of PRBC, surgical intervention or discontinuation of ECMO
  * Type 4: Any fatal bleeding

OTHER OUTCOMES:
Increase in d-dimer levels | through ECMO completion, an average of 14 days
  D-dimers level (>5000ng/ml or >50% increase in 24 h)
  * Need for transfusion of blood and blood-derived products related or not to a bleeding event
  * Coagulation parameters during the ECMO period
  * Amount of clot and fibrin visualized in the pre- and post-membrane side of the oxygenator daily (visual assessment) and after ECMO removal (assessed by a photographic quantification method).
Transfusion of blood and blood-derived products related or not to a bleeding event | through ECMO completion, an average of 14 days
  Amount of blood products transfused to patients in each groups during the course of ECMO
Coagulation parameters on ECMO | through ECMO completion, an average of 14 days
  Evaluation of fibrinogen (g/l), activated partial thromboplastin time (aPTT, seconds), prothrombin time (PT, seconds), thromboelastogram (if available), activated clotting time (ACT, seconds; if available)
Amount of clot and fibrin visualized in the pre- and post-membrane side | through ECMO completion, an average of 14 days
  Pragmatic quantification of clot visualized on both sides of the oxygenator by direct evaluation and by a photographic quantification method

CONTACTS AND LOCATIONS:
Overall Officials: Damian Ratano, MD, Principal Investigator — University Health Network, Toronto; Eddy Fan, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krueger K, Schmutz A, Zieger B, Kalbhenn J. Venovenous Extracorporeal Membrane Oxygenation With Prophylactic Subcutaneous Anticoagulation Only: An Observational Study in More Than 60 Patients. Artif Organs. 2017 Feb;41(2):186-192. doi: 10.1111/aor.12737. Epub 2016 Jun 3. PMID 27256966
- [Background] Whittlesey GC, Drucker DE, Salley SO, Smith HG, Kundu SK, Palder SB, Klein MD. ECMO without heparin: laboratory and clinical experience. J Pediatr Surg. 1991 Mar;26(3):320-4; discussion 324-5. doi: 10.1016/0022-3468(91)90510-z. PMID 2030479
- [Background] Wen PH, Chan WH, Chen YC, Chen YL, Chan CP, Lin PY. Non-heparinized ECMO serves a rescue method in a multitrauma patient combining pulmonary contusion and nonoperative internal bleeding: a case report and literature review. World J Emerg Surg. 2015 Mar 12;10:15. doi: 10.1186/s13017-015-0006-9. eCollection 2015. PMID 25774211
- [Background] Dornia C, Philipp A, Bauer S, Stroszczynski C, Schreyer AG, Muller T, Koehl GE, Lehle K. D-dimers Are a Predictor of Clot Volume Inside Membrane Oxygenators During Extracorporeal Membrane Oxygenation. Artif Organs. 2015 Sep;39(9):782-7. doi: 10.1111/aor.12460. Epub 2015 Apr 7. PMID 25845704
- [Background] Lubnow M, Philipp A, Dornia C, Schroll S, Bein T, Creutzenberg M, Diez C, Schmid C, Pfeifer M, Riegger G, Muller T, Lehle K. D-dimers as an early marker for oxygenator exchange in extracorporeal membrane oxygenation. J Crit Care. 2014 Jun;29(3):473.e1-5. doi: 10.1016/j.jcrc.2013.12.008. Epub 2013 Dec 30. PMID 24508200
- [Background] Lehle K, Philipp A, Gleich O, Holzamer A, Muller T, Bein T, Schmid C. Efficiency in extracorporeal membrane oxygenation-cellular deposits on polymethylpentene membranes increase resistance to blood flow and reduce gas exchange capacity. ASAIO J. 2008 Nov-Dec;54(6):612-7. doi: 10.1097/MAT.0b013e318186a807. PMID 19033775
- [Background] Sidebotham D, Allen SJ, McGeorge A, Ibbott N, Willcox T. Venovenous extracorporeal membrane oxygenation in adults: practical aspects of circuits, cannulae, and procedures. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):893-909. doi: 10.1053/j.jvca.2012.02.001. Epub 2012 Apr 13. No abstract available. PMID 22503344
- [Background] Lubnow M, Philipp A, Foltan M, Bull Enger T, Lunz D, Bein T, Haneya A, Schmid C, Riegger G, Muller T, Lehle K. Technical complications during veno-venous extracorporeal membrane oxygenation and their relevance predicting a system-exchange--retrospective analysis of 265 cases. PLoS One. 2014 Dec 2;9(12):e112316. doi: 10.1371/journal.pone.0112316. eCollection 2014. PMID 25464516
- [Background] Panigada M, E Iapichino G, Brioni M, Panarello G, Protti A, Grasselli G, Occhipinti G, Novembrino C, Consonni D, Arcadipane A, Gattinoni L, Pesenti A. Thromboelastography-based anticoagulation management during extracorporeal membrane oxygenation: a safety and feasibility pilot study. Ann Intensive Care. 2018 Jan 16;8(1):7. doi: 10.1186/s13613-017-0352-8. PMID 29340875